CLINICAL TRIAL: NCT06664788
Title: A Prospective, Multicenter, Randomized Clinical Investigation Evaluating the Safety and Efficacy of ETHIZIA™ Versus SURGICEL® Original in Controlling Minimal, Mild, or Moderate Soft Tissue Bleeding During Open Abdominal, Retroperitoneal, Pelvic, Thoracic (Non-cardiac) and Extremity Surgery
Brief Title: A Study of ETHIZIA Versus SURGICEL Original in Controlling Soft Tissue Bleeding During Open Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO202401; BIO202401 (Other: Ethicon,Inc)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hemostasis; Hemostatic Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ETHIZIA (Experimental): ETHIZIA will be applied at bleeding sites that meet the inclusion criteria in participants undergoing open surgery to control soft tissue bleeding. Participants will be followed up for 28 days after surgery.
  Interventions: Device: ETHIZIA
- SURGICEL Original (Active Comparator): SURGICEL Original will be applied at bleeding sites that meet the inclusion criteria in participants undergoing open surgery to control soft tissue bleeding. Participants will be followed-up for 28 days after surgery.
  Interventions: Device: SURGICEL Original

INTERVENTIONS:
Device: ETHIZIA — ETHIZIA patch will be applied to bleeding site intraoperatively.
  Arms: ETHIZIA
Device: SURGICEL Original — SURGICEL Original will be applied to bleeding site intraoperatively.
  Arms: SURGICEL Original

SUMMARY:
The objective of this clinical investigation is to evaluate the safety and efficacy of ETHIZIA to control minimal, mild, or moderate soft tissue bleeding during open surgery when compared to SURGICEL Original in the percentage of cases achieving hemostasis at 3 minutes after product application, and without re-bleeding up to 10 minutes after application.

ELIGIBILITY:
Inclusion Criteria:

Pre-operative

* Participant is scheduled to undergo an elective open, abdominal, retroperitoneal, pelvic, thoracic (non-cardiac) or extremity surgical procedure
* Participant is willing and able to give written informed consent for the clinical investigation participation

Intra-operative

* Participant in whom the Investigator can identify and visualize a target bleeding site for which any applicable conventional means for hemostasis (e.g., suture, ligature, or cautery) are ineffective or impractical
* Target Bleeding Site is identified to originate from soft tissue, defined as organ bed, loose areolar tissue, fat, lymphatic tissue/lymph node beds, and muscle
* The choice is made to use a hemostatic agent to stop the bleeding, and there is the ability to apply pressure on the surface of the hemostatic agent to achieve hemostasis
* Participant has a Target Bleeding Site with a SBSS score of 1, 2, or 3 (e.g., reflecting minimal, mild, or moderate bleeding severities)

Exclusion Criteria:

Pre-operative

* Participant is scheduled for another planned surgery within the follow-up period and the subsequent surgery would jeopardize the ETHIZIA or SURGICEL Original application
* Participant is taking multiple antithrombotic therapies in therapeutic dosage up to the time of surgery, but allowing exclusive use of acetylsalicylic acid
* Participant has an active or suspected infection at the bleeding site
* Participant is pregnant, planning on becoming pregnant, or actively breastfeeding during the 28-day follow-up period

Intra-operative

* Target bleeding site is identified to originate from parenchymal organ tissue, cardiovascular (anastomotic or cardiovascular repair sites) tissue, or is in proximity to a foramina in bone, or areas of bony confine
* Target bleeding site is from a large defect in an artery or vein that requires vascular reconstruction with maintenance of vessel patency

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Cases Achieving Hemostasis at Three Minutes Following Product Application And With No Rebleeding Up to 10 Minutes Following Application at The Target Bleeding Site | Intraoperative (up to 10 minutes)
  Cases achieving hemostasis at 3 minutes following product application & with no rebleeding up to 10 minutes following application at the target bleeding site (first bleeding site treated) will be determined by Surface Bleeding Severity Scale (SBSS). SBSS provides a clinically validated score for assessment of bleeding at the target site, and consists of 6 scores (0 = none, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, not immediately life-threatening, 5 = extreme, immediately life-threatening). A grade of 0 (None/Dry) on the SBSS is considered as achieving hemostasis.

SECONDARY OUTCOMES:
Time to Hemostasis at Target Bleeding Site | Intraoperative (up to 10 minutes)
  Time to achieve hemostasis for target bleeding site up to 10 minutes will be evaluated and presented using Kaplan-Meier estimated distribution.
Percentage of Bleeding Sites Achieving Hemostasis at Three Minutes Following Product Application And With No Rebleeding Up to 10 Minutes Following Application at All Treated Bleeding Sites | Intraoperative (up to 10 minutes)
  Percentage of bleeding sites achieving hemostasis at 3 minutes following product application & with no rebleeding up to 10 minutes following application at all bleeding sites (additional bleeding sites treated including target bleeding site) will be determined by SBSS. SBSS provides a clinically validated score for assessment of bleeding at the target site, and consists of 6 scores (0 = none, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, not immediately life-threatening, 5 = extreme, immediately life-threatening).
Time to Hemostasis for All Treated Bleeding Sites | Intraoperative (up to 10 minutes)
  Time to achieve hemostasis for all treated bleeding sites for up to 10 minutes will be evaluated.
Median Time to Hemostasis at Target Bleeding Site | Intraoperative
  Median time to hemostasis at target bleeding site will be reported.
Median Time to Hemostasis for All Treated Bleeding Sites | Intraoperative
  Median time to hemostasis for all treated bleeding sites will be reported for both groups.
Treatment Failure for Target Bleeding Site Treated and for All Treated Bleeding Sites | Intraoperative (up to 10 minutes)
  Treatment failure is defined as no hemostasis at 10 minutes or received rescue therapy prior to 10 minutes from the application of the study product.
Sustained Hemostasis at All Treated Bleeding Sites | Intraoperative
  Sustained hemostasis at all treated bleeding sites will be reported. Sustained hemostasis is defined as achieving hemostasis at 3 minutes with no rebleeding up to Day 28.
Proportion of Bleeding Sites with Rebleeding After 10 Minutes | Intraoperative
  Proportion of bleeding sites with rebleeding after 10 minutes and prior to initiation of final fascia closure will be reported. Summaries will be presented for target bleeding site and for all treated bleeding sites.
Percentage of Bleeding Sites Achieving Hemostasis with ETHIZIA or SURGICEL Original | At 30, 60, 120, 180, 240, 300, 360, 420, 480, 540, and 600 seconds
  Percentage of bleeding sites achieving hemostasis with ETHIZIA or SURGICEL Original will be reported. Summaries will be presented for target bleeding site and for all treated bleeding sites.
Proportion of Bleeding Sites Requiring More Than One Application of ETHIZIA or SURGICEL Original to Achieve Hemostasis | Intraoperative
  Proportion of bleeding sites requiring more than one application of randomized product in order to achieve hemostasis will be reported. Summaries will be presented for target bleeding site and for all treated bleeding sites.
Proportion of Bleeding Sites that Require a Second Surgical Maneuver to Achieve Hemostasis | Intraoperative
  Proportion of bleeding sites that require a second surgical maneuver (for example, adjunct product, electrocautery, etcetera) as a rescue therapy to achieve hemostasis following treatment will be reported. Summaries will be presented for target bleeding site and for all treated bleeding sites.

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon Inc. Clinical Trial, Study Director — Ethicon, Inc.
Locations (7):
- United States (6):
  - Keck Hospital of USC, Los Angeles, California
  - Washington University Barnes Jewish Hospital, St Louis, Missouri
  - Capital Health Medical Center - Hopewell, Pennington, New Jersey
  - New York Presbyterian - Weill Cornell Medical Ctr, New York, New York
  - UT Health East Texas EMS Air 1, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
- UMC Radboud, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency